CLINICAL TRIAL: NCT01356238
Title: Application of Two Different Synthetic Sequential Media for the Human IVF-ET Program
Brief Title: Application of Two Different Synthetic Sequential Media for the Human IVF-Embryo Transfer (IVF-ET) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Fertility Hospital (Other)
Responsible Party: Jeong Yoon, Maria Fertility Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MRC-1
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2009-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRC media (Experimental): Use MRC media in the human IVF-ET program
  Interventions: Other: MRC media
- Sydney IVF media (Active Comparator): Use Sydney IVF media in the human IVF-ET program
  Interventions: Other: Sydney IVF media

INTERVENTIONS:
Other: MRC media — Culture media
  Arms: MRC media
Other: Sydney IVF media — Culture media
  Arms: Sydney IVF media

SUMMARY:
Quality-controlled commercial media have been used in many in-vitro fertilization (IVF) laboratories. However, commercial media are costly and difficult to compare directly because their exact compositions are not clearly indicated. Although commercially available media have commonly been used in most IVF programs worldwide, there are several advantages to the use of in-house synthetic sequential media at IVF laboratories. First, the results of quality control should be reliable due to a stringent protocol setting-up. Second, any direct supplementations or deletions of specific components are feasible to obtain good quality embryos and high pregnancy rates since those components can be defined. Finally, dependence on commercially available media diminishes so that the laboratory can more easily accommodate unexpected situations or problems, such as a sudden increase in IVF patients. Therefore, the present study was conducted to compare the efficacy of in-house MRC media in the human IVF-embryo transfer (ET) program to that of commercially available media.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF treatment in our clinic during study period

Exclusion Criteria:

* Females older than 40 years
* Patients showed fertilization failure
* Patients with less than two 2PN embryos

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Embryo Quality | 3 Days

SECONDARY OUTCOMES:
Pregnancy and Implantation rates | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Yoon, M.S., Principal Investigator — Maria Fertility Hospital
Locations (1):
- Maria Fertility Hospital, Seoul, South Korea